CLINICAL TRIAL: NCT05217121
Title: Quadratus Lumborum Block vs Modified-Thoracolumbar Interfascial Plane Block for Pain Management After Lumbar Spinal Surgery
Brief Title: QLB vs mTLIP for Lumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 25
Record Dates: First submitted 2021-12-22; First posted 2022-02-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; Postoperative pain management; Quadratus Lumborum Block; mTLIP block
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for lumbar disc herniation surgery will be included in the study. Patients will be randomly divided into two groups (Group Q = QLB group, Group M = mTLIP group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Q = QLB group (Active Comparator): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. Tramodol will be performed for rescue analgesia.
  Interventions: Other: Quadratus Lumborum Block
- Group M = mTLIP block group (Active Comparator): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. Tramodol will be performed for rescue analgesia.
  Interventions: Other: Modified-thoracolumbar interfascial plane block

INTERVENTIONS:
Other: Quadratus Lumborum Block — The block procedure will be applied after the surgery and before extubation with patients in the prone position by using US (Vivid Q, GE Healthcare, US). Under aseptic conditions, the probe will be covered with a sterile sheath and a 22G, 80 mm block needle (Braun Stimuplex Ultra 360, Germany) will be used. After visualizing the abdominal muscles, the needle will be punctured and 5 ml of saline will be injected into the postero-lateral border of the quadratus lumborum muscle. After the block location is confirmed, 15 ml of 0.25% bupivacaine will be injected. The same process will be applied to the opposite side (30 ml totally).
  Arms: Group Q = QLB group
Other: Modified-thoracolumbar interfascial plane block — US probe will be placed vertically at the L3 vertebrae level. After visualizing the hyperechoic shadow of the spinous process and interspinous muscles as an anatomical guide point, the probe will be moved forward to the lateral to visualize the longissimus and iliocostal muscles. Between these muscles, block needle will be inserted within in plane technique in a medial-to-lateral direction in the interfascial plane. Once the needle tip will be placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 2 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 15 mL will be injected in each side (30 ml totally).
  Arms: Group M = mTLIP block group

SUMMARY:
Ultrasound-guided quadratus lumborum block (QLB) is a fascial plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle with the goal of anesthetizing the thoracolumbar nerves.

In TLIP block, local anesthetic solution is injected between the multifidus and logissimus muscles nearly at the level of the 3rd lumbar vertebra and targets the dorsal rami of the thoracolumbar nerves. Ahiskalioglu et al. defined modified-lateral technique of TLIP (mTLIP) block as a new approach. Ahiskalioglu et al. have reported that this approach has some advantages. Firstly, sonographic visualisation is more easily than the classical technique. Secondly, insertion of the needle from medial to lateral direction reduces the risk of possible neuraxial injection. It has been reported that this technique provides effective analgesia after lumbar spinal surgery.

The aim of this study is to compare US-guided mTLIP block and QLB for postoperative analgesia management after lumbar disc herniation-laminectomy surgery.

DETAILED DESCRIPTION:
Spine surgery in thoracolumbar region is one of the most common surgeries performed for the treatment of leg and back pain. Pain management is especially important for these patients since chronic pain often occurs after surgery. Severe pain may occur at postoperative period in patients following lumbar disc herniation (LDH) operation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment. US-guided interfascial plane blocks have been used increasily due to the advantages of ultrasound in anesthesia practice. Ultrasound-guided quadratus lumborum block (QLB) is a fascial plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle with the goal of anesthetizing the thoracolumbar nerves.

In TLIP block, local anesthetic solution is injected between the multifidus and logissimus muscles nearly at the level of the 3rd lumbar vertebra and targets the dorsal rami of the thoracolumbar nerves. Ahiskalioglu et al. defined modified-lateral technique of TLIP (mTLIP) block as a new approach. Ahiskalioglu et al. have reported that this approach has some advantages. Firstly, sonographic visualisation is more easily than the classical technique. Secondly, insertion of the needle from medial to lateral direction reduces the risk of possible neuraxial injection. It has been reported that this technique provides effective analgesia after lumbar spinal surgery.

The aim of this study is to compare US-guided mTLIP block and QLB for postoperative analgesia management after lumbar disc herniation-laminectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for lumbar disc herniation-laminectomy surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | Change from baseline score at postoperative 24 hour
  This scoring system includes evaluating emotional state (12 questions), physical comfort (12 questions), psychological support (7 questions), physical independence (12 questions), and pain (7 questions).

SECONDARY OUTCOMES:
The use of rescue analgesia (number of participants and rate of tramodol using) | Postoperative 24 hours period
  Tramodol using
Postoperative pain scores (NRS) | Postoperative 24 hours period
  Change from Baseline Pain Scores at Postoperative 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Ahiskalioglu A, Yayik AM, Alici HA. Ultrasound-guided lateral thoracolumbar interfascial plane (TLIP) block: Description of new modified technique. J Clin Anesth. 2017 Aug;40:62. doi: 10.1016/j.jclinane.2017.04.015. No abstract available. PMID 28625449